CLINICAL TRIAL: NCT03529071
Title: Empowering Veterans to Communicate With Healthcare Providers to Improve CKD Care
Brief Title: Empowering Veterans to Communicate With Healthcare Providers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit enough participants due to limited grant funding.
Sponsor: Northwestern University (Other)
Collaborators: Edward Hines Jr. VA Hospital (U.S. Federal Agency)
Responsible Party: Principal Investigator, Elisa Gordon, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1212869-1
Record Dates: First submitted 2018-04-20; First posted 2018-05-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Chronic Kidney Disease Stage 3
Keywords: communication; patient activation
MeSH Terms: conditions — Renal Insufficiency, Chronic; Communication; Patient Participation

STUDY DESIGN:
Intervention Model Description: Participants will be provided with a Question Prompt Sheet to use at their nephrology clinic visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CKD-Question Prompt Sheet (Experimental): Study participants will receive the CKD-QPS.
  Interventions: Behavioral: CKD-Question Prompt Sheet
- Control (No Intervention): Individuals will not receive any intervention or surveys.

INTERVENTIONS:
Behavioral: CKD-Question Prompt Sheet — The CKD-QPS is a list of 31 questions specific to CKD stage 3 patients about treatment options and self-care management designed to activate patient communication with their providers and question-asking.
  Arms: CKD-Question Prompt Sheet

SUMMARY:
The goal of this VA Innovation Seed project is to test the best approach for the delivery, feasibility, and usability of a patient-centered CKD-QPS to facilitate better Veteran understanding and engagement in their CKD-care in nephrology clinics at two geographically distinct VA hospitals (Chicago and Dallas) through on-going user feedback in real time.

DETAILED DESCRIPTION:
The goal of this VA Innovation Seed project is to test the best approach for the delivery, feasibility, and usability of a patient-centered CKD-QPS to facilitate better Veteran understanding and engagement in their CKD-care in nephrology clinics at two geographically distinct VA hospitals (Chicago and Dallas) through on-going user feedback in real time. Specifically, the pilot goals are to:

1. Test the process of delivering the CKD-QPS into clinical workflow to optimize patient and provider use of the QPS. We will rely on user (patient and provider) feedback about the feasibility of using the QPS in a real world VA environment (e.g., time required for visits using the QPS, impact on clinical workflow, patient and providers' preferences for delivering the QPS to Veterans with CKD) to adjust delivery throughout the project period.
2. Obtain continuous provider and patient feedback during the project period about QPS feasibility, use, patient participation, and provider information-giving and encouragement of question-asking during outpatient clinic visits.
3. Test how well iterative adjustments to delivery can help improve CKD-QPS patient-reported outcome measures (e.g., satisfaction with provider).

The multi-site study will take place at Hines, VA, and at VA North Texas Health System, in Dallas, TX. The intervention entails providing the CKD-Question Prompt Sheet to patients to use during patient-nephrologist (or Nurse Practitioner or Physician Assistant) clinic visits. The CKD-QPS is a 31-item list of questions about treatment options for CKD. The QPS is designed to empower patients to ask questions by reminding them of questions that they may consider asking.

Data collection entails pre-post clinic visit surveys among CKD patients, a post-clinic interview with CKD patients and nephrologists (separately), and audio-recording the clinic visit.

The knowledge gained from this study may improve other patients' satisfaction with care and communication with providers.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (age 18+) English-speaking CKD patients stage 3 (eGFR = 30-70 mL/min) who are scheduled for a clinic visit will be eligible for participation.

   1. Up to 60 will receive the QPS and all data collection activities
   2. Up to 10 will be audio recorded only
2. Nephrologists (or Nurse Practitioners or Physician Assistants) seeing CKD patients in routine clinic visits will be eligible for participation at Hines, VA.

Exclusion Criteria:

1. CKD patients who are non-English speaking, blind, hard of hearing or deaf, unable to read, and/or who are cognitively impaired will not be eligible for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Perceived efficacy in patient-physician interaction (PEPPI) | up to 2 days
  This measure, the full name of which is provided above, assesses patients' perceived self-efficacy or confidence in interacting with physicians. It includes 5 items, each of which is anchored by 1 (not at all confident) and 5 (very confident). Scores range from 5 to 25, which higher scores indicating greater confidence.

SECONDARY OUTCOMES:
# Question Prompt Sheet (QPS) Questions Asked | 1 day
  Number of questions from the QPS that were asked during the clinic encounter.
Short-form patient satisfaction questionnaire (PSQ-18) | up to 2 days
  This measure assesses patients' perceptions of satisfaction in interacting with healthcare providers.
  It includes 18 items, each of which is anchored by 1 (strongly agree) and 5 (strongly disagree). Scores range from 18 to 90, which lower scores indicating greater satisfaction with medical care.

CONTACTS AND LOCATIONS:
Overall Officials: Elisa J Gordon, PhD, MPH, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Jesse Brown Veterans Affairs Medical Center, Chicago, Illinois
  - Edward Hines, Jr. VA Hospital, Maywood, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lederer S, Fischer MJ, Gordon HS, Wadhwa A, Popli S, Gordon EJ. A question prompt sheet for adult patients with chronic kidney disease. BMC Nephrol. 2016 Oct 19;17(1):155. doi: 10.1186/s12882-016-0362-z. PMID 27760524